CLINICAL TRIAL: NCT05799534
Title: Post-COVID-19 Rehabilitation Clinics in Saudi Arabia: Improves Physical Status, Dyspnea, Fatigue, Anxiety, and Quality of Life
Brief Title: Post-Coronavirus Disease of 2019 (COVID-19) Rehabilitation Clinics in Saudi Arabia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Majmaah University (Other)
Collaborators: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Asma Alonazi, Associate Professor, Majmaah University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-472E
Record Dates: First submitted 2023-04-04; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Fatigue; Cardiopulmonary Arrest; Physical Inactivity; Muscle Weakness; Stress, Emotional; Dyspnea
Keywords: Rehabilitation; Coronavirus disease; Respiratory function; 6-min walk test; Physical Therapy
MeSH Terms: conditions — Fatigue; Heart Arrest; Sedentary Behavior; Muscle Weakness; Stress, Psychological; Dyspnea; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Before and after intervention program
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation (Experimental): The duration for 4-week, three sessions per week. Each session will last for 45-60 minutes
  Interventions: Other: Physical Therapy Rehabilitation

INTERVENTIONS:
Other: Physical Therapy Rehabilitation — Physical Therapy Rehabilitation program to to establish a novel physiotherapeutic plan to determine the effects on post-COVID-19 patients' psychoemotional condition, lung capacity, cardiorespiratory condition, and muscle strength.

SUMMARY:
This intervention study aims to evaluate the before and after changes in physical fitness, cardiorespiratory status, exercise capacity, fatigue, anxiety, dyspnea, psychoemotional conditions, and quality of life through 3 sessions per week for 4-week of an intensive therapeutic program in post coronavirus survivors. In addition, it aims to answer the main questions before and after the clinical trial study.

* Does three sessions per week for 4-week of an intensive therapeutic program improve patients' physical fitness, cardiorespiratory status, and exercise capacity?
* Does it improve physical endurance and fitness, enhancing fatigue, anxiety, and dyspnea on post coronavirus patients? Participants will ask first to answer these questionnaires before and after the intervention.
* Berg Balance Scale (BBS): to assess the patient's ability (or inability) to safely balance (standing, active, and fall risk) during a series of planned tasks.
* The Modified Medical Research Council (mMRC) Dyspnea Scale: is used to assess patients' degree of baseline functional impairment due to dyspnea from respiratory diseases.
* Depression, Anxiety, and Stress Scale- 21 Items (DASS-21): measures the emotional states of depression, anxiety, and stress.
* Fatigue Assessment Scale (FAS): evaluates symptoms of chronic fatigue.
* Quality of Life (QOL)-short form-36: to assess the quality of life and calculate eight subscales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.

After answering the questionnaires, the patients will then go through multiple tests before and after the intervention:

* A 6-min walk test (6-MWT): is the primary measure of this study to assess aerobic capacity and endurance.
* 10-meter walk test (10MWT): assess walking speed in meters per second over a short distance and assess capacity and endurance.
* Time Up and Go (TUG) test: assess lower extremity function, mobility, and fall risk. The TUG test is the shortest, most straightforward clinical balance test available to predict the risk of falls.
* 1-min sit-to-stand test (1-MSTST): assess lower extremity strength for one minute.

DETAILED DESCRIPTION:
The intervention will include all of the following exercises:

1. Breathing Exercises:

   * Breathing control:

     • Start with the breathing exercises at least twice a day, and increase to 4-6 times a day

     • Breathe in and out gently through the nose if possible.
     * If the breath is out through the mouth, the participant will instruct to purse their lips as if they are blowing out a candle
     * Attempt to release any tension in the body with each exhalation
     * Gradually try to make the breaths slower
     * Each participant will instruct to close their eyes to help focus on breathing and to relax
   * Deep breathing exercises

     * The participant will be instructed to take long, slow, and deep breaths through their nose and keep their chest and shoulders relaxed.
     * Breathe out gently and relax, like a sigh.
     * They should do three-five deep breaths.
     * Repeat for two minutes several times a day.
   * Huffing • A huff is exhaled through an open mouth and throat instead of coughing. It helps move sputum up the participants' airways so they can clear it in a controlled way.

     * To "huff," they must squeeze air quickly from their lungs through their open mouth and throat as if trying to mist up a mirror or glasses.
     * Use their abdominal muscles to assist them in squeezing out the air, but do not exert so much force that it causes wheezing or chest tightness.
     * If huffing clears their sputum, they should not need to cough. They should only cough if the sputum can clear quickly.
     * The participants should continue the breathing exercises for about 10 minutes, ideally until their chest feels clear of sputum.
2. Strengthening Exercises

   - To help restore muscle strength and increase endurance for 3 minutes daily.
   * Standing heel raise: hold on a chair, integrate arms reaching overhead when on toes. Repeat 2-3 times. Increase gradually to 8 Times (1-set)
   * Mini squats holding the chair with breathing
   * Wall push-ups hold for 8 seconds, then repetitions 2-3 times and increase to 10 repetitions.
   * For core exercises, start with 1-2 repetitions, then slowly increase to 10 repetitions.
   * Sit to stand and repeat 2-3 times. Increase gradually to 10-times
3. Mobility training or gait training

   - To increase endurance
   * Walk for at least 30 minutes without stopping five times per week
   * Start by walking on flat surfaces. As they progress and gain endurance, increase challenge by walking on hills and inclines for a 10-minute increase to 3 times a day.
   * Ascending and descending stairs with assistance if needed.
4. Home-exercise program (HEP) • All the activities above should continue at home

ELIGIBILITY:
Inclusion Criteria:

* The participants' ages from 18-45 years old
* Participants who are referred to the post-COVID clinics
* Participants who are discharged from the hospitals within 3 to 6 months ago.

Exclusion Criteria:

* If they have any active infection such as pneumonia, cardiovascular instability, pulmonary embolism, and disability or disorders.
* Musculoskeletal disorders
* Neurodegenerative diseases
* Patients unable to walk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
6-min walk test (6-MWT) | 6 minutes
  Measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Time Up and Go (TUG) test | Less 1 minute
  Measures the time needed to get up from a chair, walk 3 meters, and then return and sit back on a chair.
1-min sit-to-stand test (1-MSTST) | 1 minute
  To stand up and sit down on a chair without arm rests as many times as possible within 1 min.

SECONDARY OUTCOMES:
10-meter walk test (10MWT) | 10 minutes
  Measure used to assess walking speed in meters per second over a short distance of 14-meters.

CONTACTS AND LOCATIONS:
Overall Officials: Asma A Alonazi, DSc, Principal Investigator — Majmaah University, College of Applied Medical Sciences

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT05799534/Prot_SAP_000.pdf